CLINICAL TRIAL: NCT04100603
Title: A Non-Interventional Pilot Study to Explore the Role of Gut Flora in Clostridoides Difficile Infection
Status: Withdrawn | Type: Observational
Why Stopped: Company focus shifted
Sponsor: ProgenaBiome (Other)
Responsible Party: Sponsor
Other Study IDs: PRG-004
Record Dates: First submitted 2019-09-20; First posted 2019-09-24 (Actual); Last update posted 2025-06-05 (Actual); Status verified 2025-06

CONDITIONS: Clostridium Difficile; Clostridium Difficile Infection; Microbiome; CDI
MeSH Terms: conditions — Clostridium Infections

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Stool samples
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Patients with CDI: Patients who are infected with C. diff
  Interventions: Other: No Intervention

INTERVENTIONS:
Other: No Intervention — There is no intervention for this study

SUMMARY:
This study seeks to correlate microbiome sequencing data with information provided by patients and their medical records.

DETAILED DESCRIPTION:
The goal of this Research Study is to better understand how the genetic information in subject's microbiome correlates to infection with C. diff.

ELIGIBILITY:
Inclusion Criteria:

* Willingness to sign informed consent
* Diagnosis of C. difficile infection
* Age of 18 and older

Exclusion Criteria:

* Refusal by patient to sign informed consent form
* Treatment with antibiotics 2 weeks prior to screening
* Treatment with probiotics 6 weeks prior to screening
* History of bariatric surgery, total colectomy with ileorectal anastomosis or proctocolectomy.
* Postoperative stoma, ostomy, or ileoanal pouch
* Participation in any experimental drug protocol within the past 12 weeks
* Treatment with total parenteral nutrition
* Any clinically significant evidence of disease that could interfere with the subject's ability to enter the trial
* Inability of patient to adequately communicate with the investigator or their respective designee and/or comply with the requirements of the entire study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult patients with C. difficile infection
Sampling Method: Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2020-03-02 (Actual); Primary Completion 2030-03 (Estimated); Study Completion 2030-07-31 (Estimated)

PRIMARY OUTCOMES:
Correlation of Microbiome to Disease via Relative Abundance Found in Microbiome Sequencing | 1 year
  Relative abundance of bacterial classes within taxonomic phyla and, more broadly, within their domain will be analyzed by sequencing the gut microbiome. These data will then be categorized with C. diff infection

CONTACTS AND LOCATIONS:
Overall Officials: Sabine Hazan, MD, Principal Investigator — ProgenaBiome
Locations (1):
- ProgenaBiome, Ventura, California, United States

IPD SHARING:
Plan to Share IPD: No
Only aggregated deidentified data will be made available to other researchers.